CLINICAL TRIAL: NCT04726189
Title: A Randomized Controlled Trial on the Effect of Early Progressive Strength Exercise for Treatment of Acute Achilles Tendon Rupture. The Achilles Tendon Back-On-Track Study.
Brief Title: Early Progressive Strength Exercise for Treatment of Acute Achilles Tendon Rupture.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Christensen, PT, PHD student, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-20200041
Record Dates: First submitted 2021-01-23; First posted 2021-01-27 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Achilles Tendon Rupture
Keywords: Achilles tendon rupture; Early functional rehabilitation; Resistance training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care exercises (Active Comparator): This is the currently used treatment in the nine weeks of immobilisation with an orthosis.
  Interventions: Other: Standard exercises
- Early progressive strength exercise (Experimental): This exercise program initiates early (second week) and continues with resistance exercises with progression of the load according to individual participant toleration.
  Interventions: Other: Standard exercises plus Early progressive exercises

INTERVENTIONS:
Other: Standard exercises — Consists of a a standard exercise program with range of motion exercises from the third week and elastic band exercise from the sixth week.
  Arms: Standard care exercises
Other: Standard exercises plus Early progressive exercises — This exercise program consists of standard exercises plus the early progressive program that initiates early (second week) and continues with resistance exercises with progression of the load according to individual participant toleration. Exercises are isometric exercises from the second week and then gradually progression of load in seated heel-rise and resistance band exercises.
  Arms: Early progressive strength exercise

SUMMARY:
The purpose of this trial is to investigate the efficacy of standard care versus standard care combined with an early progressive exercise program in improving the function of the tendon and leg muscles after non-surgical treated Achilles tendon rupture

DETAILED DESCRIPTION:
Acute Achilles tendon rupture often results in long-term muscular deficits. Patients struggle to return to work and sports with high load on the lower leg. Early functional rehabilitation has shown good results, but research on resistance exercise is scarce and the reporting of the specifics of the exercises are poor.

ELIGIBILITY:
Inclusion Criteria:

* Acute total Achilles tendon rupture treated non-surgically
* Diagnosed within 3 days (of their injury)
* Age 18 - 65, able and willing to participate in the intervention
* Able to speak and understand Danish

Exclusion Criteria:

* Achilles tendon rupture close to insertion on calcaneus or in the musculo-tendinous junction of the triceps surae
* Previous Achilles tendon rupture or other conditions in either leg causing lower leg disability (pain, deficits in strength or range of movement)
* Treated with Fluoroquinolons or Corticosteroids within the last 6 months
* Diabetes or rheumatic diseases
* Severe medical illness: ASA score higher than or equal to 3. (ASA: American Society of Anesthesiologists physical status classification system)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Achilles tendon total rupture score ATRS | 13 weeks
  Validated patient reported outcome measure. It contains 10 questions about physical performance in an 11-point Likert scale from zero to ten.

SECONDARY OUTCOMES:
Achilles tendon total rupture score ATRS | Baseline, 26 and 52 weeks
  Validated patient reported outcome measure. It contains 10 questions about physical performance in an 11-point Likert scale from zero to ten.
International Physical Activity Questionnaire (IPAQ) | baseline, 13, 26 and 52 weeks
  International Physical Activity Questionnaire (IPAQ) short form Danish version. It consists of 7 items concerning physical activity as time spent performing vigorous and moderate activities, the time spent walking and sitting during the past week. The IPAQ gives an estimate of the total weekly physical activity measured in MET-minutes per week and total minutes spent sitting.(MET: The Metabolic Equivalent of Task)
Achilles tendon resting angle (ATRA) | 13 and 52 weeks
  ATRA is validated as an indirect measure of the Achilles tendon length
Achilles tendon length | 9, 13 and 52 weeks
  Ultrasound measure of achilles tendon length using Copenhagen Achilles length measure (CALM)
Isometric muscle strength | 9, 13 and 52 weeks
  maximal isometric plantar flexor muscle strength using a Fysiometer
Muscle endurance | 13 and 52 weeks
  Muscle endurance is measured in seated or standing heel-rise with MuscleLab Measurement system (Ergotest Technology, Oslo, Norway)
The fear of re-rupture | 9, 13 and 52 weeks
  The Tampa scale of Kinesiophobia (TSK) is a questionaire consisting of 17 items concerning pain and kinesiophobia and has 4 answers from "Strongly disagree" to "Strongly agree".
Adverse events | 9, 13 and 52 weeks
  The number of serious and minor adverse events is registered in a pre-defined list based on Common Terminology Criteria for Adverse Events
Compliance | 9 weeks
  The participants will register the number of exercise sessions they perform each day in a training journal.

OTHER OUTCOMES:
Cost-effectiveness outcomes | 9, 13, 26 and 52 weeks
  Work Productivity and Activity Impairment Questionnaire WPAI:GH and condition-related expenses as measured by a self-developed questionnaire
Self-reported health state | Baseline, 9, 13, 26, 52 weeks
  EQ-5D-5L is a generic health-related quality of life instrument

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Christensen, MHSc, Principal Investigator — Aalborg University Hospital, Denmark; Inge Lunding Kjær, MD, Study Chair — Aalborg University Hospital, Denmark; Jennifer A Zellers, PhD, Study Chair — Washington University School of Medicine in St. Louis, USA; Karin Grävare Silbernagel, PhD, Study Chair — University of Delaware, DE USA; Michael Skovdal Rathleff, PhD, Study Chair — Aalborg University Hospital, Denmark
Locations (2):
- Denmark (2):
  - Orthopeadic department, Physiotherapy and Occupational Therapy, Aalborg University Hospital, Aalborg
  - Orthopeadic department, Physiotherapy and Occupational Therapy, North Denmark Regional Hospital Hjørring, Hjørring

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After completion of the 1 year follow-up
Access Criteria: Researchers that provide a methodologically sound plan

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-01-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT04726189/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT04726189/SAP_001.pdf